CLINICAL TRIAL: NCT04839744
Title: A Randomized, Open-label, Parallel-Group, Comparative Study in Chinese Healthy Male Subjects to Evaluate the Safety and Pharmacokinetic Profile of TG103 Injection Produced by Two Different Manufacturing Processes
Brief Title: A Comparative Study of TG103 Produced by Two Manufacturing Processes in Chinese Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC Baike (Shandong) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSA1803-CSP-005
Record Dates: First submitted 2021-03-25; First posted 2021-04-09 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Healthy Male Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TG103 produced by the modified manufacturing process (Experimental): A single dose of TG103 (15mg) produced by the modified manufacturing process will be administered subcutaneously (SC) in healthy male subjects.
  Interventions: Drug: TG103 produced by the modified manufacturing process
- TG103 produced by the original manufacturing process original manufacturing process (Active Comparator): A single dose of TG103 (15mg) produced by the original manufacturing process will be administered subcutaneously (SC) in healthy male subjects.
  Interventions: Drug: TG103 produced by the original manufacturing process

INTERVENTIONS:
Drug: TG103 produced by the modified manufacturing process — Drug: TG103 (a modified manufacturing process), 15mg, SC
  Arms: TG103 produced by the modified manufacturing process
Drug: TG103 produced by the original manufacturing process — Drug: TG103 (the original manufacturing process), 15mg, SC
  Arms: TG103 produced by the original manufacturing process original manufacturing process

SUMMARY:
This study is designed to evaluate the comparability of TG103 injection subject to changes in the manufacturing process in Chinese healthy male subjects.

DETAILED DESCRIPTION:
This is a randomized, open-label, parallel-group, comparative study to evaluate the pharmacokinetic (PK) and pharmacodynamic (PD) profiles, safety, and immunogenicity of TG103 injection produced by two different manufacturing processes in Chinese healthy male subjects. Approximately 24 eligible subjects will be randomized in a 1:1 ratio to receive a single dose of TG103 produced by the modified manufacturing process or TG103 produced by the original manufacturing process via subcutaneous (SC) injection.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male subjects between 18 and 45 years of age, inclusive;
* 2. The subject is in good health as determined by medical history, physical examination and clinical laboratory parameters, such as vital signs, 12-lead ECG, imaging examinations (such as thyroid color Doppler ultrasound, abdominal color Doppler ultrasound, chest X-ray);
* 3. Weight ≥ 50kg, body mass index (BMI) between 19-26 kg / m2 (inclusive) [BMI = weight (kg) / height 2 (m2)];
* 4. The subject has a blood glucose between 3.9-6.1 mmol / L (exclusive) and the HbA1c < 6.5%;
* 5. From the date of signing an informed consent to at least 3 months after the administration, the subject must use reliable contraceptive methods to prevent pregnancy;
* 6. The subjects fully understand the content of the trial and the possible adverse reactions, have the ability to communicate with the researchers normally, willing and able to comply with all requirements defined in the protocol;
* 7. Voluntarily to participate in the study and sign the informed consent form.

Exclusion Criteria:

* 1. Subjects who have a history of certain allergic conditions (such as asthma, urticaria), or have a history of allergy to two or more drugs or food, or may be allergic to the test drug and the related compounds;
* 2. Have a history of serious diseases, such as neurological, hepatic, renal, cardiovascular, haematological, pulmonary diseases, or other significant diseases capable of significantly altering the absorption, metabolism, or elimination of the study drug, of constituting a risk when taking the study drug; or of interfering with the interpretation of data;
* 3. Have undergone major surgery within 3 months before screening or have severe infection within 4 weeks before screening;
* 4. With thyroid dysfunction requiring drug treatment, or not reaching clinical stability after treatment, or with other endocrine diseases that may affect blood glucose metabolism;
* 5. Have a history of or current pancreatitis (history of chronic or acute pancreatitis);
* 6. Have a history of or current cholecystitis;
* 7. With clinically significant abnormal gastric emptying (such as gastric outlet obstruction) and severe chronic gastrointestinal diseases (such as active ulcer within 6 months);
* 8. Have a history (or family history) of medullary thyroid cancer (MTC), type 2 multiple endocrine neoplasia syndrome or other hereditary diseases that are thought to induce MTC;
* 9. Have a history of malignant tumour, mental illness, depression, anxiety and epilepsy;
* 10. Have a history of drug dependence in the past one year or have a positive urine drug screen before administration;
* 11. Vaccinated within 28 days before screening or planned to be vaccinated within 1 week after receiving the study drug;
* 12. Have a positive test result of hepatitis B surface antigen, hepatitis C antibody, anti-human immunodeficiency virus antibody or anti-Treponema pallidum specific antibody;
* 13. Blood loss greater than 400 ml due to blood donation or other reasons within 3 months before screening;
* 14. Have used Glucagon-like peptide-1 (GLP-1) analogues, GLP-1 receptor agonists or any other incretin analogues three months before the planned study drug , or other drugs that are thought to affect the trial in the opinion of the researchers;
* 15. Within 3 months before administration, subjects used drugs that may cause changes in blood glucose level;
* 16. Have used any prescription drug, Chinese herbal medicine or over-the-counter drug within 15 days before screening that are capable of affecting the PK, PD and safety outcomes;
* 17. Average alcohol intake is more than 21 units of alcohol (male) per week (1 unit ≈ 360mL beer, or 45mL spirits with 40% alcohol content, or 150mL wine) within the 3 months prior to screening, or a positive ethanol breath test at screening;
* 18. Regularly consumption of caffeine is more than 600 mg per day within the 3 months prior to screening (one cup of coffee contains about 100 mg of caffeine, one cup of tea contains about 30 mg of caffeine, and one can of coke contains about 20 mg of caffeine), or those who used caffeinated products within 48 hours before administration;
* 19. Smoking more than 5 cigarettes per day within 3 months prior to screening;
* 20. According to the judgment of the researcher, the subjects have special dietary requirements;
* 21. With dermatitis or abnormal skin conditions at or around the site of administration;
* 22. Have participated in another clinical trial involving an investigational product within 3 months prior to the planned administration of the study drug; or the last dose of the previous investigational product has been given in less than 3 months before the screening; or those who would try to participate in other clinical trials during the study period;
* 23. Not suitable for this study in the researcher's opinion, such as subjects with poor compliance (long-term business trip, planned relocation, etc.).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-07-02 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Day1-5, 7,9,10, 15, and 28
Area under the plasma concentration versus time curve (AUC) | Day1-5, 7,9,10, 15, and 28

SECONDARY OUTCOMES:
Change from baseline in Fasting blood glucose(FPG) | Day1-5, and 7
  Pharmacodynamic (PD) parameters after administration of of TG103
Change from baseline in 2-hour postprandial blood glucose(2hPG) | Day1-5, and 7
  Pharmacodynamic (PD) parameters after administration of of TG103
Number of participants with treatment-emergent adverse events | Up to 28 days
  Pharmacodynamic (PD) parameters after administration of of TG103
Concentration of Antidrug antibodies(ADA) | Day1, 15, and 28
  ADA after administration of of TG103

CONTACTS AND LOCATIONS:
Overall Officials: Juan Li, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No